CLINICAL TRIAL: NCT06699758
Title: A Phase I, Single-Center, Open-Label, Dose-Escalation Clinical Trial to Assess the Safety and Tolerability of an Intranasal Memory T Lymphocytes Solution in Adult Females: vRELEASE I. (vRELEASE I)
Acronym: vRELEASE I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cristina Calvo Rey (Other)
Responsible Party: Sponsor-Investigator, Cristina Calvo Rey, Head Clinician. Pediatric and Infectious Diseases Department, Hospital Universitario La Paz
Organization: Hospital Universitario La Paz (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HULP: 6796
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-02

CONDITIONS: To Assess the Safety and Tolerability of Intranasal Administration of a Male Donor Memory T Lymphocyte Solution

STUDY DESIGN:
Intervention Model Description: Standard 3+3 dose escalation design to determine the optimal dosage of the investigational product, consisting of CD45RA- memory T lymphocytes, for intranasal administration in healthy female volunteers. The dose escalation will be based on the observed occurrence of dose-limiting toxicities (DLTs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention arm Group 1 (Experimental): Administration of a total of 3x106 cells administered over three 1x106cell doses.
  Interventions: Other: CD45RA- memory T lymphocytes cells sourced from healthy peripheral blood mononuclear cells male donors.
- Intervention arm Group 2 (Experimental): Administration of a total of 15x106 cells administered over three 5x106cell doses.
  Interventions: Other: CD45RA- memory T lymphocytes cells sourced from healthy peripheral blood mononuclear cells male donors.
- Intervention arm Group 3 (Experimental): Administration of a total of cumulative 30x106 cells administered over three 10x106cell doses.
  Interventions: Other: CD45RA- memory T lymphocytes cells sourced from healthy peripheral blood mononuclear cells male donors.

INTERVENTIONS:
Other: CD45RA- memory T lymphocytes cells sourced from healthy peripheral blood mononuclear cells male donors. — CD45RA- memory T lymphocytes cells sourced from healthy peripheral blood mononuclear cells male donors. These cells will be administered intranasally.

SUMMARY:
Proof-of-concept trial to assess the safety and tolerability of intranasal administration of a male donor memory T lymphocyte solution in females aged between 18 - 55 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects between 18 - 55 years of age.
* Participants are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Patients with the ability to comprehend and sign the informed consent.
* Written informed consent obtained prior to any screening procedures.
* Subjects in good health with no baseline disease of any kind.

Exclusion Criteria:

* Participants are not willing or able to comply with either: all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, or other study procedures.
* Participants who are currently under medical follow-up for any medical condition or who are regularly taking medication for any condition.
* Subject has experienced symptoms consistent with a respiratory infection within the 7 days prior to the administration of the investigational treatment.
* Have a known history of human immunodeficiency virus infection, Hepatitis B or Hepatitis C; testing is not required in the absence of prior documentation or known history.
* Have a known history of drug substance abuse.
* Pregnant or breastfeeding women, where pregnancy is defined as the state of a female after conception and until the termination of gestation.
* Any other condition that, in the opinion if the Investigator, may interfere with the efficacy and/or safety evaluation of the trial.
* Any condition or situation precluding or interfering with the compliance with the protocol.
* Participant is currently enrolled or has enrolled in a clinical trial three months prior to inclusion in the current study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 6 months
  Safety and tolerability will be evaluated based on the frequency and attribute of DLT (dose limiting toxicities) in the first 7 days after solution administration and the incidence of all AEs and serious adverse events (SAEs) during study period.
  The primary endpoint will be DLT, defined as any grade 3 or higher adverse event (as defined in the Common Terminology Criteria for Adverse Events (CTCAE) version 5) with an attribution of definitely or probably related to the product administration.
  The highest dose found safe in the present study will be determined as the maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
Persistence of donor cells in the nasal mucosa of participants post-administration of treatment cells | 6 months
  Persistence of donor cells in the nasal mucosa of participants post-administration of treatment cells, confirmed by the detection of male donor cells through nasopharyngeal aspirate and the presence of a Y chromosome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain